CLINICAL TRIAL: NCT03087539
Title: Exploratory Phase II Clinical Trial to Evaluate the Efficacy and Safety of Clotinab® (Abciximab) in Acute Myocardial Infarction Patients: Multicenter, Randomized, Double Blind, Placebo-controlled and Parallel Group Trial
Brief Title: Exploratory P2 Trial to Evaluate Efficacy and Safety of Clotinab® (Abciximab) in Acute MI Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ISU Abxis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ISU-CLO-201
Record Dates: First submitted 2016-09-09; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2016-07

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clotinab (Abciximab) (Experimental): 0.25 mg/kg bolus prior to PCI and then 10 ug/kg/min continuous infusion for 12 hours
  Interventions: Biological: Abciximab
- Placebo (Placebo Comparator): 0.25 mg/kg bolus prior to PCI and then 10 ug/kg/min continuous infusion for 12 hours
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Abciximab
  Other Names: Clitinab
  Arms: Clotinab (Abciximab)
Biological: Placebo
  Other Names: Plabebo
  Arms: Placebo

SUMMARY:
Exploratory Phase II Clinical Trial to Evaluate the Efficacy and Safety of Clotinab® (Abciximab) in Acute Myocardial Infarction Patients: Multicenter, Randomized, Double-Blind, Placebo-controlled and Parallel Group Trial

DETAILED DESCRIPTION:
This study was an exploratory phase 2 of Clinical Trial to evaluate the efficacy and safety of Clotinab® (Abciximab) in the acute myocardial infarction patients and was designed as a multicenter, randomized, double-blinded, placebo-controlled and parallel group study. The objective of this phase 2 clinical trial is to evaluate correlation between infarct size and major adverse cardiac event (MACE) of acute myocardial infarction patient, prearranged for percutaneous coronary intervention(PCI), to measure possibility to use infarct size as a primary efficacy test variable in phase 3 for final confirmation of safety and efficacy.

Also to determine exploratively an average variance estimation of infarct size between study drug and placebo to confirm safety and efficacy of study drug, compared to placebo and to use the estimation for calculating sample size for phase III clinical trial.

ELIGIBILITY:
Inclusion criteria

1. Patients with acute myocardial infarction having ST segment, 1 mm or above, from at least 2 consecutive segment.
2. Patients have a plan of Percutaneous Coronary Intervention (PCI)

Exclusion criteria

1. History of myocardial infarction
2. History of hypersensitivity in aspirin, heparin, or protein drugs
3. Bleeding disorders
4. Thrombocytopenia (<100,000unit/㎕)
5. Cardiogenic shock, chronic atrial fibrillation, and cancer
6. Patients with following criteria: Implanted pacemakers, defibrillators, intracranial metallic implants, pregnant, etc
7. Had a history of surgical operation within 4 weeks
8. Participated in other clinical trials within 2 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-12-14 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between the Infarct size and MACE | 18 months
  To determine correlation between infarct size and MACE

CONTACTS AND LOCATIONS:
Overall Officials: Myungho Jeong, Principal Investigator — Chonnam National Univ.
Locations (1):
- Chonnam National University, Gwangju, Chonnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
No comment